CLINICAL TRIAL: NCT04363138
Title: Link Between Eosinopenia and Bacterial Infections in the Elderly Subject Hospitalized in Geriatrics
Acronym: ELISA
Status: Completed | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00301-38
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Fever; Leukocytes; C Reactive Protein (CRP) is Less Than 20 mg/ l
Keywords: Eosinopenia; Bacterial infections
MeSH Terms: conditions — Fever; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bacterial infection: Patients with bacterial infection
- No bacterial infection: Patients without bacterial infection

SUMMARY:
The main purpose of this monocentric, non-interventional, prospective study carried out in acute geriatrics (UGA) and post-rehabilitation care, is to determine if eosinopenia is associated with bacterial infections.

DETAILED DESCRIPTION:
It's a monocentric, non-interventional, prospective study carried.

At inclusion:

Non-opposition will be collected by the investigator upon entering the Geriatric Unit.

The investigators will have all the biological and radiological results and will decide whether or not to start antibiotic treatment.

Patients will be divided into 2 groups: group with bacterial infections and the other with non-bacterial diseases.

The patient's socio-demographic data, reason for hospitalization, history, BMI, state of dependence (ADL-IADL), MMSE, treatments will be collected. Biological examinations in the phase where an infection is not suspected will also be collected (NFS, ionogram, urea, creatinemia, albumin, pre albumin, CRP, hepatocellular workup. Clinical examination during the episode may be infectious as well that biological and radiological data will be collected as well as the diagnosis made.

Antibiotic treatment is prescribed will be listed. The blood levels of eosinophils between the two groups will be compared.

Follow-up at 1 month:

The effectiveness of antibiotics will be evaluated on the absence of inflammatory syndrome and fever after the recommended antibiotic treatment and the duration of the recommended treatment. Vital status will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in Geriatrics.
* First episode of:
* Fever> 38 ° motivating the realization of a biological assessment.
* Or Leukocytes> 10 g / l and C reactive protein (CRP) > 20 mg / l.
* Be affiliated to a social security scheme.
* No oral opposition to participation in the study and use of the data.

Exclusion Criteria:

* Immunosuppression (HIV with CD4 <200 / mm3)
* Active corticosteroid therapy
* Asthma
* Chemotherapy, immunosuppressive treatment
* Malignant hematological disease, lympho or myeloproliferative syndrome
* Antibiotic therapy initiated before entering the geriatric ward
* Documented parasitosis
* Eosinophilic vasculitis
* stroke <30 days
* Patient already included in another study
* Patient under guardianship or curatorship
* Not affiliated with a social security scheme
* Oral opposition to participation in the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects above 75 years of age, hospitalized in geriatrics.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Determine if eosinopenia is associated with bacterial infections by measuring eosinophil counts. | 1 month

SECONDARY OUTCOMES:
Determine if eosinopenia is associated with the effectiveness of antibiotics by measuring eosinophil counts. | 1 month
Determine if the eosinophil counts (PNE) / neutrophil (PNN)x1000 < 4 ratio is associated with a bacterial infection by measuring this value. | 1 month
Determine if eosinopenia is associated with mortality by measuring eosinophil counts. | 1 month
Determine if deep eosinopenia is associated with bacterial involvement by measuring if this value is less than 10 per mm3. | 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle DURON, MD PhD, Study Chair — Geriatric Department, Paul Brousse Hospital
Locations (1):
- Geriatric Department, Paul Brousse Hospital, Villejuif, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mesinele L, Pujol T, Brunetti N, Neiss M, Trivalle C, Souques C, Houenou-Quenum N, Verdier S, Simon P, Vetillard AL, Houdre J, Collarino R, Mary M, Vidal JS, Kahn JE, Guichardon M, Duron E, Baudouin E. Association between low eosinophil count and acute bacterial infection, a prospective study in hospitalized older adults. BMC Geriatr. 2023 Dec 13;23(1):852. doi: 10.1186/s12877-023-04581-y. PMID 38093181